CLINICAL TRIAL: NCT01768364
Title: Antibiotic Prophylaxis When Removing Ureteric Stent After Stone Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tor Erik Sand (Other)
Responsible Party: Sponsor-Investigator, Tor Erik Sand, Professor, M.D., Ph.D., Oslo and Akershus University College
Organization: University Hospital, Akershus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012/953
Record Dates: First submitted 2013-01-14; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Ureteric Stent After Stone Surgery
MeSH Terms: interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotics (Active Comparator): will receive antibiotics
  Interventions: Drug: Trimetoprim-Sulfa (Bactrim)
- No antibiotics (Active Comparator): will not receive antibiotics
  Interventions: Other: No antibiotics

INTERVENTIONS:
Drug: Trimetoprim-Sulfa (Bactrim)
  Arms: Antibiotics
Other: No antibiotics
  Arms: No antibiotics

SUMMARY:
Is there anything to gain in giving antibiotics as prophylaxis when removing ureteric stents cystoscopically after stone surgery?

DETAILED DESCRIPTION:
Many patients undergoing stone surgery receive a ureteric stent that should be removed after 14 days. This stent is removed cystoscopically and today this is done without giving antibiotics. Some patients get urinary tract infections subject to this. However the investigators do not know how many of these patients get UTI as most are followed by their primary care doctor. With this study the investigators would like to find out whether it is possible to avoid such infections and also find out how many actually do get infected.

ELIGIBILITY:
Inclusion Criteria:

* stone surgery patients with ureteric stent that should be removed after 14 days

Exclusion Criteria:

* ongoing antibiotic treatment, allergy to trimetoprim-sulfa

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
14 days infection rate w/wo antibiotics | 14 days

SECONDARY OUTCOMES:
infection rate with ureter stent wo antibiotics | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Tor Erik Sand, MD. PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lorenskog, Lorenskog, Norway